CLINICAL TRIAL: NCT02294305
Title: Vortioxetine Versus Placebo in Major Depressive Disorder Comorbid With Social Anxiety Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Medical Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAK-S001560
Record Dates: First submitted 2014-11-11; First posted 2014-11-19 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Social Anxiety Disorder; Major Depressive Disorder
Keywords: Depression; Social Anxiety; Social Phobia; Major Depression; Vortioxetine
MeSH Terms: conditions — Phobia, Social; Depressive Disorder, Major; Depression | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vortioxetine (Experimental): Vortioxetine 10 to 20 mg PO QD for 12 weeks.
  Interventions: Drug: Vortioxetine
- Placebo (Placebo Comparator): Placebo PO QD for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine
  Other Names: Brintellix
  Arms: Vortioxetine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This placebo-controlled study is designed to determine the efficacy, safety, and tolerability of vortioxetine in the treatment of adults with Major Depressive Disorder (MDD) that is comorbid with Social Anxiety Disorder (SAD). Half of the subjects will be randomized to receive vortioxetine and the other half will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults between 18 and 70 years of age (inclusive).
2. Subjects must give written informed consent prior to any study procedures
3. Diagnosis of Major Depressive Disorder (MDD), single episode (296.2) or recurrent (296.3), according to Diagnostic and Statistical Manual of Mental Disorders, version 5 (DSM-5) criteria, as determined by psychiatric evaluation with the investigator and confirmed by the Mini-International Neuropsychiatric Interview (MINI).
4. Duration of current Major Depressive Episode must be at least 4 weeks.
5. Diagnosis of Social Anxiety Disorder (SAD) (300.23 Social Phobia) according to DSM-5 criteria, as determined by psychiatric evaluation with the Investigator and confirmed by the MINI.
6. Duration of current SAD must be at least 6 months, and SAD should be observable in subjects' lives when they are not suffering from MDD, if such periods have occurred.
7. Subjects must have a minimum total score of 60 on the Liebowitz Social Anxiety Scale (LSAS) at both Screening and Baseline visits.
8. Subjects must have a minimum total Montgomery Asberg Depression Rating Scale (MADRS) score of 20 at both Screening and Baseline visits.
9. Subjects must have a Clinical Global Inventory (CGI) Severity score of 4 or greater at both Screening and Baseline visits, where the CGI is based on a composite of MDD and SAD.
10. Male and female subjects of childbearing potential must commit to an effective form of contraception for the duration of the trial (Screening/Visit 1 through Follow-Up/Visit 10). Effective forms of contraception include: condoms with spermicide, diaphragm with spermicide, hormonal contraceptive agents (oral, transdermal, or injectable), or implantable contraceptive devices. True abstinence will also be considered an effective form of contraception.

Exclusion Criteria:

1. Subjects with any lifetime history of bipolar disorder, schizophrenia, schizoaffective disorder, Obsessive Compulsive Disorder, eating disorders, or body dysmorphic disorder. Subjects with comorbid Generalized Anxiety Disorder, dysthymia, or specific phobias can be included in the study provided that MDD and SAD are considered to be the primary clinical conditions in terms of need for treatment.
2. Subjects with substance abuse, panic disorder, or Post-Traumatic Stress Disorder, in the past 6 months before screening.
3. Subjects who started psychotherapy for SAD or MDD or had electroconvulsive therapy (ECT) in the past 6 months before screening. Subjects who have been receiving psychotherapy or Cognitive Behavioral Therapy for more than 24 weeks prior to the Baseline visit are eligible provided that the therapy continues at the same frequency for the duration of the trial.
4. Subjects who are currently pregnant or lactating, or who are of childbearing potential and not able and willing to practice an effective method of contraception (as outlined in Inclusion criterion #10) for the duration of the trial (Screening/Visit 1 through Follow-Up/Visit 10.
5. Subjects who, in the opinion of the investigator, are at a clinically significant risk for suicide. This would include prominent suicidal ideation or suicidal behavior in the past 6 months before screening.
6. Systolic blood pressure ≥165 and/or diastolic blood pressure ≥95, as measured at Screening and Baseline visits.
7. Positive Urine Drug Screen at the Screening visit, unless due to prescribed medication.
8. Any current unstable and/or clinically significant medical condition, based on history or as evidenced in screening laboratory or electrocardiogram (ECG) assessments.
9. Subjects with a history or complication of cancer or malignant tumor not in remission for at least 5 years. Basal cell skin cancers are not exclusionary.
10. Subjects receiving fluoxetine within 28 days of the Baseline visit.
11. Subjects receiving Monoamine oxidase inhibitors (MAOIs) within 14 days of the Baseline visit.
12. Subjects receiving any other psychotropic medication (including selective serotonin re-uptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), and benzodiazepines) within 14 days of the Baseline visit. Zolpidem (Ambien) PRN is allowed for insomnia if not taken more than 3 times per week for the duration of the trial.
13. Treatment refractory SAD: subjects who have a history of two or more failed treatment trials with an FDA-approved SAD treatment, each given for at least 6 weeks, during which the subject received an adequate dosage
14. Treatment refractory MDD: subjects who have a history of two or more failed treatment trials with an FDA-approved MDD treatment in the current episode

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression of Improvement (CGI-I) Responder Rate | 12 weeks
  CGI-I score of 2 (much improved) or 1 (very much improved) based on overall subject state, combining improvement in MDD and SAD features, at Visit 9/Early Termination

SECONDARY OUTCOMES:
Change in total Montgomery Asberg Depression Rating Scale (MADRS) score | Baseline and 12 Weeks
Change in total Liebowitz Social Anxiety Scale (LSAS) score | Baseline and 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Liebowitz, M.D., Principal Investigator — The Medical Research Network, LLC
Locations (1):
- The Medical Research Network, LLC, New York, New York, United States